CLINICAL TRIAL: NCT06020131
Title: Effect Of Thoracic Mobility Versus Lumbopelvic Stabilization Exercises On Lower Extremity Flexibility, Dynamic Balance And Proprioception In Patients With Chronic Ankle Instability
Brief Title: Effect Of Thoracic Mobility Versus Lumbopelvic Stabilization Exercises On Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ecemnur
Record Dates: First submitted 2023-04-30; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Chronic Ankle Instability
Keywords: chronic ankle instability; dynamic balance; proprioception; flexibility; thoracic mobility; lumbopelvic stability

STUDY DESIGN:
Intervention Model Description: The sample of study consist of patients with chronic ankle instability who gets 27 and less point from Cumberland Ankle Instability Tool. The study was conducted between November 2022 - January 2023 in Noi Physio Pilates Studio in İstanbul.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Mobility Group (Experimental): Thoracic Mobility Exercises Ankle Strengthening Home Exercises with resistive band
  Interventions: Procedure: Thoracic Mobility Rehabilitation; Procedure: Ankle Strengthening Home Exercises
- Lumbopelvic Stability Group (Experimental): Lumbopelvic stabilization exercises Ankle Strengthening Home Exercises with resistive band
  Interventions: Procedure: Lumbopelvic Stability Rehabilitation; Procedure: Ankle Strengthening Home Exercises

INTERVENTIONS:
Procedure: Thoracic Mobility Rehabilitation — Thoracic mobility exercises: Thoracic extension on foam roller, Sidelying thoracic rotation, Quadruped thoracic rotation, Squat with extension and rotation ( 10 reps x 3 set - 2 times x wk - 8 wk)
  Arms: Thoracic Mobility Group
Procedure: Lumbopelvic Stability Rehabilitation — Lumbopelvic Stabilization Exercises : Bridge with alternate leg, Single leg bridge, Four point kneeling with arm and leg extension, Side plank on front arm with knee flexed (right, left), Sitting on a Swiss Ball and hip flexion (10 reps x 3 set - 2times/wk - 8 wk)
  Arms: Lumbopelvic Stability Group
Procedure: Ankle Strengthening Home Exercises — Ankle Strengthening exercises with resistive band (dorsiflexion, plantarflexion, inversion, eversion) (10 reps x 3 set - 3 times/wk)

SUMMARY:
The aim of the study is to investigate the effectiveness of thoracic mobility versus lumbopelvic stabilization exercises combined with ankle strengthening exercises with resistive band on patients with chronic ankle instability in terms of lower extremity flexibility, proprioception and dynamic balance.The participants were divided into two group as Thoracic Mobility group (n=15) and Lumbopelvic Stability group (n=15). In addition their exercise programs (2 times/wk, 8 wk duration), both groups were given home exercise ankle strengthening exercises.(3 sets/ 10 reps, 3 times/wk.)

DETAILED DESCRIPTION:
The aim of the study is to investigate the effectiveness of thoracic mobility versus lumbopelvic stabilization exercises combined with ankle strengthening exercises with resistive band on patients with chronic ankle instability in terms of lower extremity flexibility, proprioception and dynamic balance. The study were conducted in Noi Physio Pilates Studio in Istanbul between November 2022 - January 2023 during 8 weeks. 30 volunteers with chronic ankle instability were included according to Cumberland Ankle Instability Tool (CAIT). The cut off value for the CAIT test was determined as 27. Participants who received 27 or less than this value were included in the study. All participants were right dominant. Lower extremity flexibility was assessed with Active Straight Leg Raise Test, proprioception (hip, knee, ankle) was assessed with Joint Position Sense Test using electronic goniometer. Determined angles for joints; hip flexion angle as 75°, knee flexion angle as 50° and ankle dorsiflexion as 10° plantarflexion as 40°.Y Balance Test (anterior, posterolateral, posteromedial) was used for evaluating dynamic balance. 30 participants were divided into two groups as thoracic mobility and lumbopelvic stability group. Both groups were given ankle strengthening exercises (dorsiflexion, plantarflexion, inversion and eversion) with resistive band. Home exercises were performed 3 days a week for a total of 3 sets of 10 repetitions. Thoracic mobility group was given; thoracic extension on foam roller, sidelying thoracic rotation, quadruped thoracic rotation, squat with extension and rotation. Lumbopelvic stabilization group was prescribed; bridge with alternate leg, single leg bridge, four point kneeling with arm and leg extension, side plank on front arm with knee flexed (right, left), sitting on a Swiss Ball and hip flexion.Sessions took approximately 50 minutes and exercise program was planned twice a week for 8 weeks, 16 sessions total. Both groups were given ankle strengthening exercises (dorsiflexion, plantarflexion, inversion and eversion) with resistive band. Home exercises were performed 3 days a week for a total of 3 sets of 10 repetitions.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years
* Having at least two previous lateral ankle sprain of same ankle.
* At least one episode of "giving way" wtihin previous 6 months.
* Having persistent symptoms during functional activities and being free of.
* Symptoms from any previous lower limb injuries.
* No other lower extremity injuries.

Exclusion Criteria:

* Having any systemic illness (eg. Rheumatoid arthritis, DM).
* Any surgery history related to fractures or disorders.
* Getting steroid injection or physiotherapy intervention previous 6 months.
* Being a pregnant and existence of tumor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) | 8 weeks
  CAIT is questionnaire' has 9 items with scores ranging from 0 to 30, with lower scores indicating worse stability

SECONDARY OUTCOMES:
Active Straight Leg Raise Test | 8 weeks
  It is used for evaluation of lower extremity flexibility.
Y Balance Test | 8 weeks
  Dynamic balance test for right and left leg including three directions (anterior, posterolateral, posteromedial)
Joint Position Sense Test | 8 weeks
  It is a test for measuring proprioception of joints. (Hip, knee, ankle)

CONTACTS AND LOCATIONS:
Overall Officials: Ecem Nur TAKINDI, MSc, Principal Investigator — Yeditepe University, Institute of Health Science, Sports Physiotherapy Department; Elif Tuğçe ÇİL, PhD, Study Director — Yeditepe University, Institute of Health Science, Sports Physiotherapy Department
Locations (1):
- Noi Physio Pilates Studio, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants were included to study accorcing to Informed Consent Form (ICF). Datas and informations were recorded.
Supporting Information: ICF
Time Frame: 8 week
Access Criteria: Informed consent form was used for gathering demographic information from participants. Cumberland Ankle Instability Tool (CAIT) was used for assesing chronic ankle instability. Cut off value was determined as ≤27 points.

REFERENCES:
- [Background] Herzog MM, Kerr ZY, Marshall SW, Wikstrom EA. Epidemiology of Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):603-610. doi: 10.4085/1062-6050-447-17. Epub 2019 May 28. PMID 31135209
- [Background] Al-Mohrej OA, Al-Kenani NS. Chronic ankle instability: Current perspectives. Avicenna J Med. 2016 Oct-Dec;6(4):103-108. doi: 10.4103/2231-0770.191446. PMID 27843798
- [Background] Hertel J, Corbett RO. An Updated Model of Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):572-588. doi: 10.4085/1062-6050-344-18. Epub 2019 Jun 4. PMID 31162943
- [Background] Kobayashi T, Gamada K. Lateral Ankle Sprain and Chronic Ankle Instability: A Critical Review. Foot Ankle Spec. 2014 Aug 1;7(4):298-326. doi: 10.1177/1938640014539813. Epub 2014 Jun 24. PMID 24962695
- [Background] Hiller CE, Kilbreath SL, Refshauge KM. Chronic ankle instability: evolution of the model. J Athl Train. 2011 Mar-Apr;46(2):133-41. doi: 10.4085/1062-6050-46.2.133. PMID 21391798
- [Background] Chen ET, Borg-Stein J, McInnis KC. Ankle Sprains: Evaluation, Rehabilitation, and Prevention. Curr Sports Med Rep. 2019 Jun;18(6):217-223. doi: 10.1249/JSR.0000000000000603. PMID 31385837
- [Background] Vuurberg G, Hoorntje A, Wink LM, van der Doelen BFW, van den Bekerom MP, Dekker R, van Dijk CN, Krips R, Loogman MCM, Ridderikhof ML, Smithuis FF, Stufkens SAS, Verhagen EALM, de Bie RA, Kerkhoffs GMMJ. Diagnosis, treatment and prevention of ankle sprains: update of an evidence-based clinical guideline. Br J Sports Med. 2018 Aug;52(15):956. doi: 10.1136/bjsports-2017-098106. Epub 2018 Mar 7. PMID 29514819
- [Background] Cleland JA, Mintken PE, McDevitt A, Bieniek ML, Carpenter KJ, Kulp K, Whitman JM. Manual physical therapy and exercise versus supervised home exercise in the management of patients with inversion ankle sprain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2013;43(7):443-55. doi: 10.2519/jospt.2013.4792. Epub 2013 Apr 29. PMID 23628755
- [Background] Czajka CM, Tran E, Cai AN, DiPreta JA. Ankle sprains and instability. Med Clin North Am. 2014 Mar;98(2):313-29. doi: 10.1016/j.mcna.2013.11.003. Epub 2014 Jan 10. PMID 24559877
- [Background] Needle AR, Tinsley JE, Cash JJ, Koeval BK, Barton JA, Howard JS. The effects of neuromuscular electrical stimulation to the ankle pronators on neural excitability & functional status in patients with chronic ankle instability. Phys Ther Sport. 2023 Mar;60:1-8. doi: 10.1016/j.ptsp.2022.12.001. Epub 2022 Dec 9. PMID 36634453
- [Background] Hall EA, Docherty CL, Simon J, Kingma JJ, Klossner JC. Strength-training protocols to improve deficits in participants with chronic ankle instability: a randomized controlled trial. J Athl Train. 2015 Jan;50(1):36-44. doi: 10.4085/1062-6050-49.3.71. Epub 2014 Nov 3. PMID 25365134
- [Background] Donovan L, Hertel J. A new paradigm for rehabilitation of patients with chronic ankle instability. Phys Sportsmed. 2012 Nov;40(4):41-51. doi: 10.3810/psm.2012.11.1987. PMID 23306414
- [Background] Rodriguez-Merchan EC. Chronic ankle instability: diagnosis and treatment. Arch Orthop Trauma Surg. 2012 Feb;132(2):211-9. doi: 10.1007/s00402-011-1421-3. Epub 2011 Nov 5. PMID 22057817
- [Background] Molla-Casanova S, Ingles M, Serra-Ano P. Effects of balance training on functionality, ankle instability, and dynamic balance outcomes in people with chronic ankle instability: Systematic review and meta-analysis. Clin Rehabil. 2021 Dec;35(12):1694-1709. doi: 10.1177/02692155211022009. Epub 2021 May 31. PMID 34058832
- [Background] Xue X, Tao W, Xu X, Jin Z, Li Q, Wang Y, Gu X, Wang R, Hua Y. Do exercise therapies restore the deficits of joint position sense in patients with chronic ankle instability? A systematic review and meta-analysis. Sports Med Health Sci. 2023 Jan 23;5(1):67-73. doi: 10.1016/j.smhs.2023.01.001. eCollection 2023 Mar. PMID 36994176
- [Background] Kosik KB, McCann RS, Terada M, Gribble PA. Therapeutic interventions for improving self-reported function in patients with chronic ankle instability: a systematic review. Br J Sports Med. 2017 Jan;51(2):105-112. doi: 10.1136/bjsports-2016-096534. Epub 2016 Nov 2. PMID 27806951
- [Background] McCann RS, Crossett ID, Terada M, Kosik KB, Bolding BA, Gribble PA. Hip strength and star excursion balance test deficits of patients with chronic ankle instability. J Sci Med Sport. 2017 Nov;20(11):992-996. doi: 10.1016/j.jsams.2017.05.005. Epub 2017 May 25. PMID 28595864
- [Background] Sciascia A, Cromwell R. Kinetic chain rehabilitation: a theoretical framework. Rehabil Res Pract. 2012;2012:853037. doi: 10.1155/2012/853037. Epub 2012 May 14. PMID 22666599
- [Background] Lee J-I, Kim T-H. Effects of hip joint strengthening exercises and lumbopelvic stabilization exercises on balance and instability of adults with functional ankle instability. International Journal of Human Movement and Sports Sciences. 2021;9(4):757-764. doi:10.13189/saj.2021.090421
- [Background] Terada M, Pietrosimone BG, Gribble PA. Alterations in neuromuscular control at the knee in individuals with chronic ankle instability. J Athl Train. 2014 Sep-Oct;49(5):599-607. doi: 10.4085/1062-6050-49.3.28. Epub 2014 Aug 21. PMID 25144597
- [Background] Khalaj N, Vicenzino B, Heales LJ, Smith MD. Is chronic ankle instability associated with impaired muscle strength? Ankle, knee and hip muscle strength in individuals with chronic ankle instability: a systematic review with meta-analysis. Br J Sports Med. 2020 Jul;54(14):839-847. doi: 10.1136/bjsports-2018-100070. Epub 2020 Jan 14. PMID 31937576
- [Background] Jeong H-J, Kim B-J. The effect of thoracic joint mobilization on the changes of the thoracic kyphosis angle and static and dynamic balance. Biomedical Science Letters. 2019;25(2):149-158. doi:10.15616/bsl.2019.25.2.149
- [Background] Cruz-Diaz D, Lomas-Vega R, Osuna-Perez MC, Contreras FH, Martinez-Amat A. Effects of 6 Weeks of Balance Training on Chronic Ankle Instability in Athletes: A Randomized Controlled Trial. Int J Sports Med. 2015 Aug;36(9):754-60. doi: 10.1055/s-0034-1398645. Epub 2015 May 13. PMID 25969966
- [Background] Karartı C, Bilgin S, Büyükturan Ö, Büyükturan B, Dadalı Y, Bek N. Lumbopelvi̇k Motor Kontrol, postüral Denge ve Fiziksel Performans Arasındaki İlişki. Türk Fizyoterapi ve Rehabilitasyon Dergisi. 2019. doi:10.21653/tfrd.425735
- [Background] Vuurberg G, Kluit L, van Dijk CN. The Cumberland Ankle Instability Tool (CAIT) in the Dutch population with and without complaints of ankle instability. Knee Surg Sports Traumatol Arthrosc. 2018 Mar;26(3):882-891. doi: 10.1007/s00167-016-4350-4. Epub 2016 Oct 6. PMID 27714439
- [Background] Lee DK, Kang MH, Lee TS, Oh JS. Relationships among the Y balance test, Berg Balance Scale, and lower limb strength in middle-aged and older females. Braz J Phys Ther. 2015 May-Jun;19(3):227-34. doi: 10.1590/bjpt-rbf.2014.0096. Epub 2015 May 29. PMID 26039033
- [Background] Liebenson C, Karpowicz AM, Brown SH, Howarth SJ, McGill SM. The active straight leg raise test and lumbar spine stability. PM R. 2009 Jun;1(6):530-5. doi: 10.1016/j.pmrj.2009.03.007. PMID 19627942
- [Background] Olsson L, Lund H, Henriksen M, Rogind H, Bliddal H, Danneskiold-Samsøe B. Test-retest reliability of a knee joint position sense measurement method in sitting and prone position. Advances in Physiotherapy. 2004;6(1):37-47. doi:10.1080/14038190310009894
- [Background] McCann RS, Johnson K, Suttmiller AMB. Lumbopelvic Stability and Trunk Muscle Contractility of Individuals with Chronic Ankle Instability. Int J Sports Phys Ther. 2021 Jun 2;16(3):741-748. doi: 10.26603/001c.22132. PMID 34123527
- [Background] Boucher JA, Preuss R, Henry SM, Dumas JP, Lariviere C. The effects of an 8-week stabilization exercise program on lumbar movement sense in patients with low back pain. BMC Musculoskelet Disord. 2016 Jan 14;17:23. doi: 10.1186/s12891-016-0875-4. PMID 26762185
- [Background] Alahmari KA, Kakaraparthi VN, Reddy RS, Silvian P, Tedla JS, Rengaramanujam K, Ahmad I. Combined Effects of Strengthening and Proprioceptive Training on Stability, Balance, and Proprioception Among Subjects with Chronic Ankle Instability in Different Age Groups: Evaluation of Clinical Outcome Measures. Indian J Orthop. 2020 Jul 15;55(Suppl 1):199-208. doi: 10.1007/s43465-020-00192-6. eCollection 2021 May. PMID 34122771
- [Background] Anguish B, Sandrey MA. Two 4-Week Balance-Training Programs for Chronic Ankle Instability. J Athl Train. 2018 Jul;53(7):662-671. doi: 10.4085/1062-6050-555-16. PMID 30192681
- [Background] Tamura A, Shimura K, Inoue Y. Hip flexibility and dynamic balance ability in soccer players with functional ankle instability. Trauma Care. 2021;1(3):206-214. doi:10.3390/traumacare1030018
- [Background] Tahoon A, Shendy, S, El-khozamy, H, Baky, WA. Flexibility deficit in chronic ankle instability. Case Medical Research. 2019. doi:10.31525/ct1-nct04083391
- [Background] Brolinson PG, Rogers M, Edison J. Functional and kinetic chain evaluation of the hip and pelvis. The Hip and Pelvis in Sports Medicine and Primary Care. 2016:37-64. doi:10.1007/978-3-319-42788-1_3
- [Background] Myer GD, Chu DA, Brent JL, Hewett TE. Trunk and hip control neuromuscular training for the prevention of knee joint injury. Clin Sports Med. 2008 Jul;27(3):425-48, ix. doi: 10.1016/j.csm.2008.02.006. PMID 18503876